CLINICAL TRIAL: NCT03458182
Title: Recalled Exertional Breathlessness and Improved Predicted Exercise Capacity: A Randomized Controlled Trial
Brief Title: Breathlessness During Exercise: Experience and Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Magnus Ekström (Other)
Responsible Party: Sponsor-Investigator, Magnus Ekström, MD, PhD, Associate Professor, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECALL18
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Dyspnea; Breathlessness
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Added exercise (Experimental): After completion of the standard exercise test, an intervention period of 2 minutes of low intensity exercise is added.
  Interventions: Other: Added exercise
- No intervention (No Intervention): No added exercise period (normal exercise test).

INTERVENTIONS:
Other: Added exercise — After completion of the standard exercise test, an intervention period of 2 minutes of low intensity exercise is added.
  Arms: Added exercise

SUMMARY:
Breathlessness during exertion is a major limiting factor for patients' physical capacity and activity. Increased exertional breathlessness often results in impaired activity, spiraling deconditioning and further worsening of exertional breathlessness, quality of life and prognosis.

Recalled symptoms (from memory) can differ substantially from the actually experienced symptoms.The recall of symptom intensity is affected by several factors including the experienced peak intensity and the intensity at the end of the episode. This 'Peak-end-rule' has been reported in studies of pain, and in breathlessness in daily life and during exercise. A randomized trial reported that adding a time period with decreased pain at the end of a colonoscopy decreased the patient's recalled total pain of the event, improved their overall perception of the event and made them more willing to participate in similar procedures in the future.

Pulmonary rehabilitation training is the first line treatment for exertional breathlessness and deconditioning in cardiorespiratory disease. However, the training as well as physical activities of daily life are often limited by the person's perception of his/her capacity, which is based on recalled breathlessness during exertion. The person's predicted breathlessness - that is, the level of breathlessness that the person predicts will occur during a future activity, is likely a major determinant of his/her willingness to participate in training as well as of the level of physical activity in daily life.

To improve the effectiveness of cardio-pulmonary rehabilitation training and the patients' health status, new approaches for decreasing the perceived exertional breathlessness and optimize training are needed.

The investigators hypothesize that adding a period of lower breathlessness intensity at the end of training might be a way to manipulate the recalled (remembered) symptom intensity during the training, and to improve the subject's perceived future exercise capacity and willingness to participate in physical exercise/ training.

DETAILED DESCRIPTION:
The primary purpose is to test whether adding a period of lower level of exertional breathlessness at the end of an exercise test decreases the overall level of recalled breathlessness for the test.

Secondly the investigators aim to evaluate factors that affect the level of recalled breathlessness, and whether decreased exertional breathlessness results in the participant's reporting lower predicted future exertional breathlessness and higher exercise capacity.

Information about the study and the pre-test questionnaire will be sent home to patients referred for standard cycle exercise testing. The pre-test questionnaire is completed by the participant at home or before the exercise test. Eligibility is confirmed and written informed consent is obtained for all participants by the investigator before starting the exercise test. All patients included in the RCT (randomized clinical trial), randomizations, and patients included in the observational sub-study are registered in a log file including study ID, Swedish identification number and test date, stored securely at the Department of Clinical Physiology.

Standard exercise test is performed according to clinical practice, current international guidelines and guidelines from the Swedish association for Clinical Physiology. Testing is done on bicycle ergometers with small incremental increases in workload every minute. The level of breathlessness is self-reported by the participant each 2 minutes on a modified Borg CR10 (mBorg) scale between 0 (none) and 10 (maximal). The level of perceived exertion is self-reported by the participant on the Borg RPE (rating of perceived exertion) scale between 7 (none) and 20 (maximal), and standard parameters of exercise testing are measured according to clinical routine practice.

At the end of the regular exercise test conducted according to clinical practice, with the participant still on the test cycle, a sealed opaque envelope is broken by the staff with a code that randomly allocates the participant in a 1:1 ratio to either an additional 2 minutes of low intensity exercise testing (intervention group), or to no additional testing (control group). During the intervention period. The workload used will be about 50% of the maximal workload but lowered if needed, and assessments are conducted including of breathlessness, perceived exertion, breathing frequency and blood pressure. A period of a few minutes of lower exertion ('cool down') at the end of the exercise test is clinical practice in many laboratories including in the USA, and is not expected to affect the safety or diagnostic properties of the exercise test. As an added precaution the investigators have obtained opinions from well-known experts in cardiac stress testing (Dr. Olle Pahlm and Dr. Paul Kligfield). In additions to this ST loops will also be used to further enhance the diagnostic properties of the test. ST loops are not currently used by default in the study laboratory.

A post-test questionnaire is completed by the participant 30-90 min after the exercise test.

Patients completing the exercise test who fulfill the inclusion criteria and give their written informed consent are included in an observational longitudinal follow-up study. The study data are cross-linked with medical records and governmental public registries regarding diagnoses, procedures and hospitalizations (National Patient Register) and mortality (Causes of Death Register) with up to 10 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Persons referred and eligible for standard exercise stress testing
* Able to read, write and understand sufficient Swedish to participate

Exclusion Criteria:

* Duration of exercise test ≤ 3 minutes
* Maximal breathlessness intensity ≤ 3/10 during the test
* Clinical or cardiovascular instability during the exercise test before randomization as judged by the investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Recalled breathlessness | Post-test questionnaire completed by the participant 30-90 min after the exercise test.
  Recalled overall intensity of breathlessness (0-10 mBorg scale) during the exercise test.

SECONDARY OUTCOMES:
Predicted future exertional breathlessness | Post-test questionnaire completed by the participant 30-90 min after the exercise test.
  Predicted future exertional breathlessness (0-10 mBorg scale.
Predicted future exercise capacity | Post-test questionnaire completed by the participant 30-90 min after the exercise test.
  Predicted future exercise capacity (7-20 Borg scale).
Recalled peak breathlessness intensity during the exercise test | Post-test questionnaire is completed by the participant 30-90 min after the exercise test.
  Recalled peak intensity of breathlessness (0-10 mBorg scale).
Factors influencing the difference between experienced and recalled breathlessness of the exercise test | Post-test questionnaire is completed by the participant 30-90 min after the exercise test.
  Recalled descriptors
Recalled descriptors of breathlessness and their intensity | Post-test questionnaire is completed by the participant 30-90 min after the exercise test.
  Recalled descriptors of breathlessness and their intensity
Recalled overall and peak level of exertion during the exercise test | Post-test questionnaire is completed by the participant 30-90 min after the exercise test.
  Recalled overall and peak level of exertion (7-20 mBorg scale).
Overall perception of the exercise test | Post-test questionnaire is completed by the participant 30-90 min after the exercise test.
  Recalled descriptors
Diagnoses (IHD; heart failure; pulmonary disease; other) during 10 years follow-up | 10 year follow-up
  Swedish National Patient Register
Rate of revascularization and coronary bypass operation during 10 years follow-up | 10 year follow-up
  Swedish National Patient Register
Rate of hospitalization (overall and as for diagnosis) during 10 years follow-up | 10 year follow-up
  Swedish National Patient Register
Rate of mortality and causes of death (overall and as for diagnosis) during 10 years follow-up | 10 year follow-up
  Swedish Causes of Death Register

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Ekström, MD,PhD, Study Director — Lund University
Locations (1):
- Blekingesjukhuset, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Redelmeier DA, Katz J, Kahneman D. Memories of colonoscopy: a randomized trial. Pain. 2003 Jul;104(1-2):187-94. doi: 10.1016/s0304-3959(03)00003-4. PMID 12855328
- [Background] Kahneman D. Experienced Utility and Objective Happiness: A Moment-Based Approach. In: D. Kahneman and A. Tversky (Eds.) Choices, Values and Frames. New York: Cambridge University Press and the Russell Sage Foundation 2000.
- [Background] Meek PM, Lareau SC, Anderson D. Memory for symptoms in COPD patients: how accurate are their reports? Eur Respir J. 2001 Sep;18(3):474-81. doi: 10.1183/09031936.01.00083501. PMID 11589344
- [Background] Stulbarg MS, Carrieri-Kohlman V, Gormley JM, Tsang A, Paul S. Accuracy of recall of dyspnea after exercise training sessions. J Cardiopulm Rehabil. 1999 Jul-Aug;19(4):242-8. doi: 10.1097/00008483-199907000-00005. PMID 10453431
- [Background] Bolton CE, Bevan-Smith EF, Blakey JD, Crowe P, Elkin SL, Garrod R, Greening NJ, Heslop K, Hull JH, Man WD, Morgan MD, Proud D, Roberts CM, Sewell L, Singh SJ, Walker PP, Walmsley S; British Thoracic Society Pulmonary Rehabilitation Guideline Development Group; British Thoracic Society Standards of Care Committee. British Thoracic Society guideline on pulmonary rehabilitation in adults. Thorax. 2013 Sep;68 Suppl 2:ii1-30. doi: 10.1136/thoraxjnl-2013-203808. No abstract available. PMID 23880483
- [Background] Puente-Maestu L, Palange P, Casaburi R, Laveneziana P, Maltais F, Neder JA, O'Donnell DE, Onorati P, Porszasz J, Rabinovich R, Rossiter HB, Singh S, Troosters T, Ward S. Use of exercise testing in the evaluation of interventional efficacy: an official ERS statement. Eur Respir J. 2016 Feb;47(2):429-60. doi: 10.1183/13993003.00745-2015. Epub 2016 Jan 21. PMID 26797036
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Brudin L, Jorfeldt L, Pahlm O. Comparison of two commonly used reference materials for exercise bicycle tests with a Swedish clinical database of patients with normal outcome. Clin Physiol Funct Imaging. 2014 Jul;34(4):297-307. doi: 10.1111/cpf.12097. Epub 2013 Oct 31. PMID 24171936
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Hareendran A, Leidy NK, Monz BU, Winnette R, Becker K, Mahler DA. Proposing a standardized method for evaluating patient report of the intensity of dyspnea during exercise testing in COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:345-55. doi: 10.2147/COPD.S29571. Epub 2012 May 28. PMID 22745534
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Williams M, Garrard A, Cafarella P, Petkov J, Frith P. Quality of recalled dyspnoea is different from exercise-induced dyspnoea: an experimental study. Aust J Physiother. 2009;55(3):177-83. doi: 10.1016/s0004-9514(09)70078-9. PMID 19681739
- [Background] Banzett RB, O'Donnell CR, Guilfoyle TE, Parshall MB, Schwartzstein RM, Meek PM, Gracely RH, Lansing RW. Multidimensional Dyspnea Profile: an instrument for clinical and laboratory research. Eur Respir J. 2015 Jun;45(6):1681-91. doi: 10.1183/09031936.00038914. Epub 2015 Mar 18. PMID 25792641
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441